CLINICAL TRIAL: NCT02883322
Title: Adaptation Process of Patient-Reported Outcomes, an eVALuation Study
Acronym: APPROVALS
Status: Completed | Type: Observational
Sponsor: GUILLEMIN Francis, MD (Other)
Collaborators: Societe Francaise de Rhumatologie (Other); Région Lorraine (Unknown)
Responsible Party: Sponsor-Investigator, GUILLEMIN Francis, MD, Médecin coordinateur de module, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: APPROVALS
Record Dates: First submitted 2016-08-19; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Initial: Patients answering the initial translation
  Interventions: Other: Cross cultural adaptation of patient reported outcomes (PRO)
- Committee-only: Patients answering the translation modified by an expert committee
  Interventions: Other: Cross cultural adaptation of patient reported outcomes (PRO)
- BT-only: Patients answering the translation modified with the use of a back-translation
  Interventions: Other: Cross cultural adaptation of patient reported outcomes (PRO)
- Both: Patients answering the translation modified by an expert committee with the use of a back-translation
  Interventions: Other: Cross cultural adaptation of patient reported outcomes (PRO)

INTERVENTIONS:
Other: Cross cultural adaptation of patient reported outcomes (PRO) — Process used to adapt a questionnaire from one cultural setting to another

SUMMARY:
Objectives: To identify the respective contributions of back-translations and of the expert committee in the process of cultural adaptation of patient reported outcome with an experimental design in the adaptation process :

Four translations of a questionnaire will be produced:

* A simple translation by two translators, who serves as the basis for the three other translations
* A translation made with the use of a back-translation.
* A translation with review by an expert committee.
* A translation the use of a back-translation and review by an expert committee.

Properties of each translation will be analyzed and compared

ELIGIBILITY:
Inclusion Criteria:

* Adult (other 18 years)
* Able to read, understand and answer the adapted questionnaire
* Having a medical condition targeted by the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a chronic condition, susceptible to answer the adapted questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
heiQ questionnaire | baseline
  Face/content validity, reliability, structural validity

CONTACTS AND LOCATIONS:
Overall Officials: Francis Guillemin, MD, PHD, Study Director — Inserm, CHRU Nancy, Université de Lorraine, CIC 1433 Épidémiologie Clinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein J, Santo RM, Guillemin F. A review of guidelines for cross-cultural adaptation of questionnaires could not bring out a consensus. J Clin Epidemiol. 2015 Apr;68(4):435-41. doi: 10.1016/j.jclinepi.2014.11.021. Epub 2014 Dec 17. PMID 25698408
- [Result] Epstein J, Osborne RH, Elsworth GR, Beaton DE, Guillemin F. Cross-cultural adaptation of the Health Education Impact Questionnaire: experimental study showed expert committee, not back-translation, added value. J Clin Epidemiol. 2015 Apr;68(4):360-9. doi: 10.1016/j.jclinepi.2013.07.013. Epub 2013 Sep 29. PMID 24084448